CLINICAL TRIAL: NCT00103467
Title: A Phase 1 Trial to Evaluate the Safety and Immunogenicity of an Anthrax Recombinant Protective Antigen Vaccine
Brief Title: Trial to Evaluate the Safety and Immunogenicity of an Anthrax Recombinant Protective Antigen Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VaxGen (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VAX005
Record Dates: First submitted 2005-02-08; First posted 2005-02-09 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-02

CONDITIONS: Prevention of Anthrax Infection

INTERVENTIONS:
Biological: rPA102 Vaccine

SUMMARY:
The purpose of this phase 1 study is to evaluate the safety and immunogenicity of rPA102 vaccine, using anthrax vaccine adsorbed (AVA) as a comparator.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the study and give written informed consent. A signed informed consent must be in place before the initiation of any study interventions.
* Healthy male or female aged 18 to 40 years old (inclusive) without significant physical or clinical laboratory abnormalities.
* Two intact upper arms with sufficient intramuscular (IM) tissue in the deltoid region for vaccine administration.
* For females, negative serum pregnancy test at screening and agreement to use adequate birth control during the first 3 months of the study.
* Willingness and ability to return for all follow-up visits and blood draws for the duration of the study.
* Willingness to complete the Volunteer Diary and to report concomitant medications and adverse events (AEs) to the study site monitors during the study period.

Exclusion Criteria:

* Prior history of, or known exposure to any form of B. anthracis or any anthrax immunization.
* Member of the Armed Services (Active Duty or Reserve) since 1990, with history of previous anthrax vaccination.
* Employment in an industry involved in contact with ruminant animals, veterinary sciences, or other exposure to B. anthracis.
* Expected to be noncompliant with study visits or planning to move within 8 months.
* Body mass index of >35 or <19.
* Known allergy to aluminum hydroxide, formaldehyde, benzethonium chloride, latex, kanamycin, or any other aminoglycoside antibiotics (such as gentamycin).
* Pregnancy (positive urine pregnancy test within 24 hours prior to vaccination), or lactation.
* HIV positive (by history or screening ELISA).
* Hepatitis B or C positive (by history or screening HBsAg/anti-HCV ELISA).
* Active or past internal organ, hematologic malignancy, or metastatic cutaneous malignancy.
* History of, or current autoimmune disease, including but not limited to systemic lupus erythematosus, scleroderma, and polyarteritis.
* Immunodeficiency or unstable medical condition as determined by baseline medical history, physical exam, and laboratory assessment.
* Received, or plans to receive, licensed live vaccines within 30 days of study vaccination.
* Received, or plans to receive, licensed killed vaccines within 14 days of study vaccination.
* Received, or plans to receive, immunoglobulin or other blood products within 60 days of study vaccination.
* Received, or plans to receive, experimental drugs/vaccines within 30 days of study vaccination.
* Received, or plans to receive, systemic immunosuppresive therapy, radiation therapy, or high-dose inhaled steroids within 30 days of study vaccination.
* Use of systemic chemotherapy within 5 years prior to study.
* History of Guillain-Barre Syndrome.
* In addition to the conditions listed above, the following may qualify as a reason to exclude a volunteer from the study: fever along with moderate or serious illness within 3 days of vaccination or any condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the study evaluations. Pending resolution of these symptoms, a volunteer may be reconsidered for vaccination.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100
Dates: Start 2003-06

PRIMARY OUTCOMES:
Safety and immunogenicity of 3 doses over 4 different dose ranges.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Emory University School of Medicine, Atlanta, Georgia
  - Dept. of International Health - Johns Hopkins University Bloomberg School of Public Health, Baltimore, Maryland
  - St. Louis University - SoLutions/SLUtest, St Louis, Missouri
  - Baylor College of Medicine, Houston, Texas